CLINICAL TRIAL: NCT03619226
Title: Evaluation of the Ability of Newly Developed Adhesives to Absorb Moisture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP284_1
Record Dates: First submitted 2018-07-13; First posted 2018-08-07 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Stoma Ileostomy
MeSH Terms: interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test patch (Experimental): two adhesive patches are applied to the abdominal area
  Interventions: Other: test patch

INTERVENTIONS:
Other: test patch — the test patch consists of an adhesive patch

SUMMARY:
The aim of this evaluation is to investigate the ability of newly developed adhesive patches to absorb moisture.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have intact skin on the area used in the evaluation
4. Have an abdominal area accessible for application of test product (assessed by investigator)
5. Negative pregnancy test for fertile women
6. Signed document claiming use of safe contraceptives for fertile women

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemo-therapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigator)
5. Participating in interventional clinical investigations or have previously participated in this evaluation. Exception: Participation in other Coloplast sponsored clinical investigations or evaluations is accepted under the circumstances that the subject has paused the activities in the investigation/evaluation and are otherwise complying with the inclusion and exclusion criteria of this (CP284) Evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, Principal Investigator — Head of the pre-clinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Patch (Adhesive Patch With Sensor System) + Hard Physical Activities + Normal Daily Activities: Two adhesive patches are applied to the abdominal area on two consecutive days. The first patch is worn with normal daily activities and the second patch is stress tested during half an hour spinning activities in humid environment plus normal day activities.
Period: Overall Study
Arm/Group | Test Patch (Adhesive Patch With Sensor System) + Hard Physical Activities + Normal Daily Activities
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteers
Arm/Group | Test Patch
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Resistance (Moisture in the Adhesive)
Description: The outcome measure is described as number of events where the sensor system reacted to a false positive leak.
  Moisture in adhesive is measured using a sensor system. Moisture influences the resistance of the sensor system. Intense moisture/sweat does not result in false positive leak signals. The signal response to moisture/sweat is different to the response to leaks.
Time Frame: 3 days
Population: Healthy volunteers
Measure: Number; unit: Number of false positive leaks
Groups:
- Test Patch (Adhesive Patch With Sensor System) + Normal Daily Activities; Test Patch (Adhesive Patch With Sensor System) + Hard Physical Activities + Normal Daily Activities: two adhesive patches are applied to the abdominal area on two consecutive days. The first patch is worn with normal daily activities and the second patch is stress tested during half an hour spinning activities in humid environment plus normal day activities.
Arm/Group | Test Patch (Adhesive Patch With Sensor System) + Normal Daily Activities | Test Patch (Adhesive Patch With Sensor System) + Hard Physical Activities + Normal Daily Activities
Number analyzed (Participants) | 6 | 6
Number of false positive leaks | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 days
Description: [Not specified]
Arm/Group | Test Patch (Adhesive Patch With Sensor System) + Hard Physical Activities + Normal Daily Activities
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT03619226/Prot_SAP_000.pdf